CLINICAL TRIAL: NCT07368296
Title: Impact of Lingual Attachment Placement on White Spot Lesion Development in Clear Aligner Orthodontic Patients : A Randomized Controlled Clinical Trial
Brief Title: Impact of Lingual Attachment on WSL Development in Clear Aligner Patients: A Randomized Controlled Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JUST20240550
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: White Spot Lesion of Tooth
Keywords: Lingual attachments; Buccal attachments; White spot lesions; Quantitative light induced fluorescence; Clear aligner therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lingual attachment participants (Active Comparator): In this group composite attachments were placed on the lingual/palatal surfaces of teeth for clear aligner therapy
  Interventions: Other: Lingual attachment participants
- Buccal attachment participants (Active Comparator): In this group composite attachments were placed on the buccal surfaces of teeth for clear aligner therapy
  Interventions: Other: Lingual attachment participants

INTERVENTIONS:
Other: Lingual attachment participants — WSL were measured on tooth surfaces of orthodontic patients wearing clear aligners with lingual attachments

SUMMARY:
White spot lesions (WSLs) are a common esthetic complication during orthodontic treatment. While clear aligners (CAs) generally reduce WSL risk compared to fixed appliances, composite attachments remain plaque-retentive sites. This two-arm clinical trial investigated the effect of shifting attachments to lingual surfaces on WSL development.

DETAILED DESCRIPTION:
A randomized controlled trial was conducted on 52 patients (18-35 years) undergoing CA therapy. Participants were allocated to two groups (n=26) for each: conventional buccal attachments (control) and lingual/palatal attachments (intervention). WSLs and plaque were assessed at baseline (T0) and six months (T1) using quantitative light-induced fluorescence (QLF). Outcomes included lesion area (pixels), mean fluorescence loss (ΔF), maximum depth (ΔFmax), and plaque index (ΔR30). Statistical analysis employed paired and independent t-tests, chi-square, and multivariable regression (α<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Medically fit young adults
* The patient should have mild to moderate crowding or spacing of teeth.
* The treatment plan should be non-extraction.
* Patients should have optimum oral hygiene before beginning the treatment.
* The patient may have a maximum of three teeth with either fillings or dental prostheses.

(According to the British national institute of health, NIH 2016).

Exclusion Criteria:

* Patients with defective enamel, generalized enamel disorder, or extensive dental restorations.
* Patients with syndromes or orofacial anomalies.
* Patients with salivary gland diseases or taking medications that may affect oral flora or salivary functions.
* Patients who are pregnant or diabetic.
* Patients use mouth rinses or any extra form of fluoride other than toothpaste.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
White spot lesion area | Before treatment and after 6 months
  Lesion area measured in pixels
Delta F | Before treatment and after 6 months
  Loss of fluorescence which reflects loss in minerals
Delta F max | Before treatment and after 6 months
  Measures the deepest point of the lesion

SECONDARY OUTCOMES:
Plaque measurement | Before treatment and after 6 months
  It measures the amount of plaque on tooth surfaces

CONTACTS AND LOCATIONS:
Locations (1):
- postgraduate orthodontic clinics at JUST, Irbid, Jordan